CLINICAL TRIAL: NCT05088395
Title: Analysis of Circulating Tumor mArkers in Blood 4 - ALCINA 4
Acronym: ALCINA4
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IC 2020-11
Record Dates: First submitted 2021-09-28; First posted 2021-10-21 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Cancer
Keywords: circulating biomarkers; Cohort
MeSH Terms: conditions — Neoplasms | interventions — Blood Specimen Collection; Biopsy

STUDY DESIGN:
Intervention Model Description: Interventional study (blood collections and possibly tumor sample collection depending on cohort type) on single group cohorts (each cohort is defined in the arms below).
  Detection study of blood tumor biomarkers and correlation with clinicopathological characteristics.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (10):
- Cohort 1: "SENOLOC" (Other): Detecting residual disease after surgery is absolutely crucial in oncology, as this detection could allow the personalisation of post-operative treatments based on the presence of residual disease.
  The laboratory wishes to develop a new technique for the detection of circulating tumour DNA, based on the recognition of translocation fragments in circulating DNA by shallow whole genome sequencing. This is an original approach, which to our knowledge has not been tested so far with the envisaged bioinformatics approach and could potentially be more sensitive than the techniques currently used to detect residual disease after surgical removal of localised (non-metastatic) breast cancer.
  The analysis will therefore focus on the search for tumour chromosomal translocations, which will need to be differentiated from possible germline chromosomal translocations. The collection of constitutional DNA is therefore planned in this cohort.
  Interventions: Other: Blood sample
- Cohort 2: "Immuno-TNBC " (Other): The aim for this cohort is to study the role that variations in circulating tumour DNA might have as a marker associated with response during chemoimmunotherapy.
  A fresh biopsy (subsequently stored frozen) is required for mutational profiling analysis (which will be used to track circulating tumour DNA in the blood). In addition, it will be used to analyse currently recognised biological tissue factors of response to chemoimmunotherapy (PD-L1 labelling, mutational load, ...) and to identify possible associations with circulating tumour DNA variations.
  Constitutional DNA analysis is necessary for the determination of point mutations present in the tumour (to be differentiated from polymorphisms present at the constitutional level), as the determination of these mutations is essential to monitor circulating tumour DNA and will therefore be collected.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 3: "Trans-TNBC" (Other): The objective of this cohort is the development of new plasma tests, for example based on the detection of chromosomal translocations of circulating tumor DNA.
  The hypothesis is that these tests would allow the detection of relapse, the prediction of treatment efficacy and the monitoring of treatment efficacy at different stages of cancer in patients with triple-negative breast cancer, either in the non-metastatic phase with planned neo-adjuvant treatment, or in the metastatic phase. The number of inclusions between these 2 populations (neo-adjuvant and metastatic) will be monitored at the operational level to avoid an excessive imbalance towards one group.
  Interventions: Other: Blood sample
- Cohort 4: "Treg" (Other): The purpose of this cohort, based on the previous results, is to:
  1. quantify the expression level of target genes on tumor Regulatory T (Tregs) at the protein level,
  2. perform multiparametric FACS analysis on blood and tumor samples from patients treated at the Institut Curie, with breast or ovary cancer and to understand the potential of these targets as biomarkers of disease.
  In the context of this ALCINA-4 cohort n°4, for breast and ovary patients, 40 ml of blood will be collected and tumor fragments obtained from surgery (50 breast patients) or therapeutically required biopsy (30 ovary patients). No additional biopsy than the ones belonging to the therapeutic process will be performed in this protocol. Biopsies performed as part of standard of care will be used if sufficient material is available.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 5: "Pembro Neo" (Other): The purpose of this cohort is to determine the detection rate of circulating tumour DNA (ctDNA) before and after surgery in the blood of patients who received neoadjuvant treatment with chemoimmunotherapy for early triple-negative breast cancer (TNBC).
  There will be two subgroups : patients who have not yet started neoadjuvant treatment (subcohort 1) and patients who have already started neoadjuvant treatment (subcohort 2).
  Biopsy of a tumour lesion will be performed before the start of neoadjuvant treatment (only for subcohort 1). The collection of constitutional DNA, plasma and circulating tumour DNA are planned in this cohort at different time points.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 6: "THL" (Other): The main objective of this exploratory cohort is to characterize the detection rate of ctDNA before and during therapy with T-DXd (Trastuzumab deruxtecan) for patients with HER2-low metastatic breast cancer, requiring treatment with T-DXd.
  Tumor biopsy will be performed after inclusion and before the start of treatment on cycle 1 day 1 for at least 30 patients. The collection of constitutional DNA, is planned in this cohort at different time points : T1 and T2 (before treatment start) are critical to evaluate the intra-patient reproducibility of liquid biomarkers. T3 will investigate the response to therapy while T4 will focus on resistance mechanisms.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 7:"CDK4/6 adjuvant" (Other): The purpose of this cohort is to determine the prognostic impact of circulating tumor DNA detection and monitoring in patients receiving a CDK4/6 inhibitor in adjuvant breast cancer.
  50 ml of blood will be collected in EDTA tubes for constitutional DNA and plasma for research of circulating biomarkers at different time points (4 time points).
  Interventions: Other: Blood sample
- Cohort 8:"ctDNA adjuvant " (Other): The purpose of this cohort is to estimate the incidence of ctDNA detection in patients with early-stage breast cancer during follow-up to detect metastatic relapse earlier in asymptomatic patients.
  ctDNA analysis will be performed using various techniques, including next-generation sequencing (NGS), with or without analysis of tumor tissue, taken as part of the standard care.
  40 ml of blood samples will be collected at four time points:
  * enrollment,
  * 6 months (+/- 15 days),
  * 12 months (+/- 15 days),
  * 18 months (+/- 15 days) after inclusion.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 9:"ADN-CIRC-Poumon " (Other): The purpose of this cohort is to:
  * Generate data on the levels and nature of circulating tumor DNA under chemo-immunotherapy.
  * Monitor the evolution of the circulating immune response under systemic chemo-immunotherapy.
  Tumor biopsy will be performed after inclusion and before the start of treatment.
  50 ml of blood samples will be collected at four time points:
  * At inclusion, before starting neoadjuvant treatment
  * At the start of cycle 3 (C3J1) of neoadjuvant treatment
  * At the time of surgery (after neoadjuvant treatment)
  * At the start of monitoring, i.e. 3 months (+/- 1 month) after surgery.
  Interventions: Other: Blood sample; Other: Biopsy
- Cohort 10: "UM TENEO" (Other): The purpose of this cohort is to :
  * Evaluate recurrence-free survival (RFS) after R0/R1 surgery
  * Assess effectiveness of Tebentafusp associated with surgery for patients with uveal melanoma metastases.
    3 sub-cohorts :
  * Sub-cohort 1: HLA-A*02:01-positive patients, eligible for R0 surgery and Tebentafusp (n=20)
  * Sub-cohort 2: HLA-A*02:01-negative patients, eligible for R0 surgery and immunotherapy at next relapse (n=20)
  * Sub-cohort 3: HLA-A*02:01 positive patients, not eligible for R0 surgery but eligible for Tebentafusp (n=20).
  Tumor biopsy will be performed during surgery (sub-cohorts n°1 and 2) or after inclusion (sub-cohort n°3).
  40 ml of blood will be collected in EDTA tubes for constitutional DNA and circulating DNA in plasma for research of biomarkers at 4 time points.
  Interventions: Other: Blood sample; Other: Biopsy

INTERVENTIONS:
Other: Blood sample — Depending on the clinical context studied and the biomarkers studied and/or sought, the timing of blood samples will vary between cohorts. There may be up to 4 samples taken per patient for up to 24 months.
Other: Biopsy — If a specific tumor sample is required, it will be collected only once during the study
  Arms: Cohort 10: "UM TENEO"; Cohort 2: "Immuno-TNBC "; Cohort 4: "Treg"; Cohort 5: "Pembro Neo"; Cohort 6: "THL"; Cohort 8:"ctDNA adjuvant "; Cohort 9:"ADN-CIRC-Poumon "

SUMMARY:
Multi-cohort exploratory prospective study. Participation in the ALCINA 4 study does not change the standard management of the patient, including the treatments administered. A sampling schedule will be set up for each cohort.

Depending on the clinical context studied and the biomarkers studied and/or sought, the timing of blood samples will vary between cohorts. There may be up to 4 samples taken per patient for up to 12 or 18 months. If a specific tumor sample is required, it will be collected only once during the study.

DETAILED DESCRIPTION:
The ALCINA 4 study is a prospective biological cohort study based on the analysis of circulating tumour biomarkers obtained by blood sampling, with comparison - if necessary - with tumour material obtained by biopsy.

Circulating tumour biomarkers in blood have been the subject of much research for several decades, leading to the development in the 1980s of serum protein markers still in use today (CA15.3, ACE, CA125...). In the last decade, research has focused on circulating tumour cells (CTCs), circulating endothelial cells (CECs) and more recently on the detection of circulating tumour DNA (ctDNA) and exosomes (or microvesicles). While ctDNA seems to have a very promising future, other circulating elements such as microRNA are also part of what can/will be studied from a simple blood sample. Broadly speaking, the potential clinical interests of these circulating biomarkers are :

* diagnostic (diagnosis of cancer, or especially diagnosis of genetic mutations present in a known cancer)
* prognostic (to adapt the intensity of treatment to the expected outcome of the patient)
* predictive of the efficacy of targeted therapies (according to the mutational profile of the cancer)
* to study mechanisms of resistance during treatment . The multiplicity of these potential blood biomarkers is matched by a large number of detection techniques, for example for CTCs or ctDNA.

The major new challenge in research on circulating biomarkers is to replace molecular analyses on tumour tissue obtained by biopsy (e.g. the search for somatic cancer mutations) by a simple blood sample ("liquid biopsy"). This objective, which is technologically possible in the very short term and particularly interesting - both medically (for patients) and economically - requires the comparison of data from blood markers with those from tumour tissue samples. Furthermore, there is an important trend to combine several levels of analysis together (e.g. ctDNA and serum protein markers) to refine the performance of blood tests.

ELIGIBILITY:
Inclusion Criteria:

* Patient treated for cancer at one of the participating center
* 18 years old or higher
* Signed informed consent form
* Patient not deprived of their liberty or under guardianship (including temporary guardianship)
* Patient covered by social security scheme
* Patient with no compliance issue (related to geographical, social or psychological reasons) for study follow up
* Other additional criteria will be defined (defining tumor type and clinical setting), by cohort

If a biopsy tumor sample is to be taken:

* Tumor considered as accessible by biopsy (at the investigator's discretion).
* Normal blood coagulation tests (if applicable, and in case of a non-superficial tumor lesion).
* No anticoagulant or antiaggregant treatment for the biopsy.

Exclusion Criteria :

Pregnant and/or breast-feeding women depending on cohort.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2050 (Estimated)
Dates: Start 2022-05-19 (Actual); Primary Completion 2031-06-01 (Estimated); Study Completion 2031-06-01 (Estimated)

PRIMARY OUTCOMES:
Detection rate of circulating biomarkers in cohort 1 | Baseline
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 2 | Baseline
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 2 | Before treatment
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 2 | At 3 weeks of treatment
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 2 | At 9 weeks of treatment
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 2 | At disease progression
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 1 | Before surgery
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 1 | After surgery (from 3 to 5 weeks)
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 1 | After surgery (from 2 to 3 months)
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 3 | Baseline
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 3 | At the end of cycle 1 (each cycle is 21 days)
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 3 | After surgery (from 2 to 3 months)
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 3 | At disease progression
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 4 | At pre-surgery or before starting treatment
  Positivity rate of the detection technique (in %)
Detection rate of circulating biomarkers in cohort 4 | At 6 weeks after surgery or after start of treatment
  Positivity rate of the detection technique (in %)

CONTACTS AND LOCATIONS:
Overall Officials: Francois-Clement BIDARD, Principal Investigator — Institut Curie
Locations (2):
- France (2):
  - Institut Curie, Paris
  - Institut Curie, Saint-Cloud

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets. Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).